CLINICAL TRIAL: NCT04436263
Title: Investigation of in Vivo Anti-inflammatory and Anti-platelet Mechanisms of Natural Extract by Modulating PAF Metabolism and Actions
Brief Title: Cardioprotective Properties of Natural Anti-Platelet Activating Factor Extract From Winery By-products in Healthy Women
Acronym: NAPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Elizabeth Fragopoulou, Assistant Professor in Biological Chemistry, Harokopio University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HarokopioU_anti-PAF extract
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Platelet Aggregation and Inflammation
Keywords: winery by-products; natural extract; postprandial study; platelet aggregation; anti-inflammatory; healthy women; Platelet-activating factor
MeSH Terms: conditions — Inflammation | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement (Experimental): Ethanol-water extract of winery by-products
  Interventions: Behavioral: Supplement
- Placebo (Placebo Comparator): Maltodextrin-based placebo
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Supplement — A sufficient quantity of the winery by-products will be extracted on an industrial scale and capsules will be produced, each one containing 110mg of phenolic compounds (gallic acid equivalents).Volunteers will consume 6 capsules along with a standardized meal (1131 kcal, 19.7% carbohydrates, 11.2% protein, 66.7% fat) and blood will be drown before the meal consumption and at specific time points for the next 6h
  Arms: Supplement
Behavioral: Placebo — A look-alike placebo containing maltodextrin will be prepared.Volunteers will consume 6 capsules along with a standardized meal (1131 kcal, 19.7% carbohydrates, 11.2% protein, 66.7% fat) and blood will be drown before the meal consumption and at specific time points for the next 6h
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the anti-platelet and anti-inflammatory properties of a winery by-products extract as well as to detect extract compounds and their metabolites in biological fluids. The study is a randomized, double-blind, crossover, placebo controlled postprandial study in healthy women.

DETAILED DESCRIPTION:
The well-known cardioprotective and metabolic effects of wine consumption are mainly attributed to its micro-constituents. Grape pomace (GP) is a by-product of the winemaking process and consists mainly of skins and seeds. Winery by-products are a cheap and rich source of similar-to wine micro-constituents, which can be used either to enrich other foods or to be included in food supplements targeting the prevention or partially the therapy of cardiovascular diseases.In this line, our previous results revealed the potent in vitro anti-platelet effects of a specific ethanol-water extract rich in Platelet-Activating Factor inhibitors from winery by-products.

The purpose of this study is to investigate the in vivo anti-platelet and anti-inflammatory properties of the specific winery by-products extract as well as to detect the extract compounds and their metabolites in biological fluids.

Therefore a randomized double-blind, crossover, placebo controlled postprandial study in healthy women will be implemented. For this purpose, 15 healthy women will participate in the protocol. The two daily trials will take place during specific days based on their menstrual cycle. Three days before each blood collection the volunteers will be instructed to abstain from food and beverages rich in phenolic compounds and their dietary intake will be recorded (three 24h recalls and one food frequency questionnaire). The blood collections will be carried out after 8h fasting. At trial day, the volunteers will bring the first morning urine sample and anthropometric measurements will take place (weight, height, waist/hip circumference, bioelectrical impedance). Then a venous catheter will be placed and after 10 minutes the fasting blood will be collected. Volunteers will proceed to the consumption of a standardized meal (1131 kcal, 19.7% carbohydrates, 11.2% protein, 66.7% fat) along with the capsules (study extract or placebo). The type of the capsules consumed (study extract or placebo) will be randomized and blind during the two intervention days for both volunteers and investigators. Blood will be drown after the meal consumption and for the next 6h (every 30minutes for the first 4h and every 1h for the next 2h). Serum, plasma, platelet-rich plasma, leukocyte-rich plasma and urine samples will be isolated at certain time points during trial days so that the anti-platelet, anti-inflammatory and antioxidant effects of the study extract can be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Females
* BMI: 22-32 kg/m2

Exclusion Criteria:

* Systematic medication
* Chronic disease conditions
* Specific dietary conditions (vegeterian, vegan...)
* Eating disorders

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-06-20 (Estimated); Study Completion 2021-06-20 (Estimated)

PRIMARY OUTCOMES:
Effect on platelet aggregation | Change between timepoints (before meal consumption, 30min, 90min, 150min, 210min, 300min) of the 6hour trial and between the two different interventions
  % Change of EC50 value of platelet aggregation against PAF
Effect on platelet aggregation | Change between timepoints (before meal consumption, 30min, 90min, 150min, 210min, 300min) of the 6hour trial and between the two different interventions
  % Change of EC50 value of platelet aggregation against ADP
Effect on platelet aggregation | Change between timepoints (before meal consumption, 30min, 90min, 150min, 210min, 300min) of the 6hour trial and between the two different interventions
  % Change of EC50 value of platelet aggregation against Collagen
Effect on inflammatory markers | Change between timepoints (before meal consumption, 60min, 120min, 180min, 210min, 240min, 300min, 360min) of the 6hour trial and between the two different interventions
  Change in PAF biosynthetic enzymes activity (lyso-PAF AT)
Effect on inflammatory markers | Change between timepoints (before meal consumption, 60min, 120min, 180min, 210min, 240min, 300min, 360min) of the 6hour trial and between the two different interventions
  Change in PAF biosynthetic enzymes activity (PAF-CPT)
Effect on inflammatory markers | Change between timepoints (before meal consumption, 60min, 120min, 180min, 240min, 360min) of the 6hour trial and between the two different interventions
  Change in PAF levels Change in PAF degradation enzyme activity (Lp-PLA2) Change in PAF levels IL6
Effect on inflammatory markers | Change between timepoints (before meal consumption, 0min, 30min, 60min, 90min, 120min, 150min, 180min, 210min, 240min, 300min, 360min) of the 6hour trial and between the two different interventions
  Change in PAF degradation enzyme activity (Lp-PLA2)
Effect on inflammatory markers | Change between timepoints (before meal consumption, 0min, 30min, 60min, 90min, 120min, 150min, 180min, 210min, 240min, 300min, 360min) of the 6hour trial and between the two different interventions
  IL-6

SECONDARY OUTCOMES:
Effect on classical biochemical markers | Change between timepoints (before meal consumption, 0min, 30min, 60min, 90min, 120min, 150min, 180min, 210min, 240min, 300min, 360min) of the 6hour trial and between the two different interventions
  Total serum cholesterol
Effect on classical biochemical markers | Change between timepoints (before meal consumption, 0min, 30min, 60min, 90min, 120min, 150min, 180min, 210min, 240min, 300min, 360min) of the 6hour trial and between the two different interventions
  LDL-cholesterol
Effect on classical biochemical markers | Change between timepoints (before meal consumption, 0min, 30min, 60min, 90min, 120min, 150min, 180min, 210min, 240min, 300min, 360min) of the 6hour trial and between the two different interventions
  HDL-cholesterol
Effect on classical biochemical markers | Change between timepoints (before meal consumption, 0min, 30min, 60min, 90min, 120min, 150min, 180min, 210min, 240min, 300min, 360min) of the 6hour trial and between the two different interventions
  TAG
Effect on classical biochemical markers | Change between timepoints (before meal consumption, 0min, 30min, 60min, 90min, 120min, 150min, 180min, 210min, 240min, 300min, 360min) of the 6hour trial and between the two different interventions
  uric acid
Effect on classical biochemical markers | Change between timepoints (before meal consumption, 0min, 30min, 60min, 90min, 120min, 150min, 180min, 210min, 240min, 300min, 360min) of the 6hour trial and between the two different interventions
  Glucose
Effect on classical biochemical markers | Change between timepoints (before meal consumption, 0min, 30min, 60min, 90min, 120min, 150min, 180min, 210min, 240min, 300min, 360min) of the 6hour trial and between the two different interventions
  Insulin
Detection and estimation of extract compounds metabolites | Change between timepoints (before meal consumption, 60min, 120min, 240min, 360min) of the 6hour trial and between the two different interventions

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition-Dietetics, Harokopio University, Athens, Greece

IPD SHARING:
Plan to Share IPD: No